CLINICAL TRIAL: NCT02357797
Title: Adjunctive Vortioxetine in Schizophrenia
Acronym: AVIS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Christoph U. Correll, MD, Professor of Psychiatry, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-645
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia; Negative Symptoms
MeSH Terms: conditions — Schizophrenia | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vortioxetine (Active Comparator): Vortioxetine will be initiated at 10 mg / day for 1 month, followed by 20 mg /day for the remainder of the trial. The dose of vortioxetine can be lowered to 10 mg for tolerability reasons.
  Interventions: Drug: Vortioxetine
- Placebo (Placebo Comparator): Matching placebo pills will be initiated at 10 mg / day for 1 month, followed by 20 mg /day for the remainder of the trial. The dose of placebo can be lowered to 10 mg for tolerability reasons.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vortioxetine
  Other Names: Brintellix
  Arms: Vortioxetine
Other: Placebo
  Arms: Placebo

SUMMARY:
This is a 16-week, randomized, double-blind, parallel group, placebo-controlled study comparing adjunctive vortioxetine with identically appearing adjunctive placebo pills in 88 stable patients with a research diagnosis of schizophrenia determined with the Structured Clinical Interview for DSM (SCID). Patient randomization will be stratified by illness duration (i.e., </=5 years and >5 years) in order to allow for post-hoc analyses examining whether earlier illness moderates greater negative and /or cognitive symptom reduction in response to vortioxetine.

DETAILED DESCRIPTION:
This is a 16-week, randomized, double-blind, parallel group, placebo-controlled study comparing adjunctive vortioxetine with identically appearing adjunctive placebo pills in 88 stable patients with a research diagnosis of schizophrenia determined with the Structured Clinical Interview for DSM (SCID). Patient randomization will be stratified by illness duration (i.e., </=5 years and >5 years) in order to allow for post-hoc analyses examining whether earlier illness moderates greater negative and /or cognitive symptom reduction in response to vortioxetine.

Patients with clinical stability for at least 3 months and stable antipsychotic and psychotropic medication treatment for at least the last 4 weeks and without relevant depression, positive psychotic symptoms or extrapyramidal symptoms EPS will be eligible. After written informed consent, patients will undergo a screening visit to confirm full study eligibility. If all in- and exclusion criteria are fulfilled, patients will undergo a baseline assessment and then be randomized 1:1 to 16 weeks of adjunctive treatment with vortioxetine or placebo. Subsequently, patients will be seen at week 1, 2, 4 and monthly for the next 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient
2. SCID diagnosis of schizophrenia
3. Age 18-65 years old
4. Treated with an adequate dose of one or a maximum of two antipsychotic medications for at least 3 months, with a stable dose for at least the last 4 weeks, and willing to continue for up to 16 weeks.
5. No antidepressant treatment for at least 8 weeks prior to randomization.
6. Treatment with other concomitant, non-antipsychotic, psychiatric medications is allowed, but must be unchanged for at least 8 weeks, with a stable dose for at least the last 4 weeks, and willing to continue for 16 weeks. Benzodiazepines must not be given within 8 hours of the cognitive assessment. Treatment with non-psychiatric medications is unrestricted.
7. PANSS Negative subscore >14 with at least two of the items at a level >/=4 (moderate)
8. PANSS Positive subscore </=14 with not more than one of the items at a level >/=4 (moderate) for patients who have been stable outpatients for <1 year. A PANSS Positive subscore of </=18 is acceptable for patients who have been stable outpatients for >/=1year and whose psychotic symptoms do not affect behavior in a clinically relevant way as per investigator assessment. - . In order to avoid simple double counting, any rating on P1 ("delusions") will not be considered as an additional symptom for determination of eligibility based on PANSS positive subscore when a specific delusion is present that is rated either on P5 ("grandiosity") or P6 ("suspiciousness/paranoia"), whereas delusions not captured by P5 ("grandiosity") or P6 ("suspiciousness/paranoia"), will be rated under P1 ("delusions") and counted toward the sum score used to determine study eligibility).
9. HAMD-17 total score </=12
10. Simpson Angus Score of any item <3
11. English-speaking
12. Competent and willing to sign informed consent

Exclusion Criteria:

1. Structural brain disease
2. Mental retardation by history and estimated IQ <70 (WRAT-III Word Reading)
3. Autism-spectrum disorder diagnosis by history
4. Any serious chronic medical illnesses that in the view of the investigator will interfere with the patient's ability to comply with the study procedures or that will interfere with cognition.
5. Active substance abuse or dependence in the past 8 weeks
6. Intolerance to or inefficacy of vortioxetine in the past
7. Acute anger to self or others as per investigator assessment
8. Pregnant or breastfeeding females
9. Unwilling or unable to be sexually abstinent or not using an effective form of birth control if they are sexually active
10. Current treatment with a Monoamine Oxidase Inhibitor (MAOI)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2016-02; Primary Completion 2023-10-01 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Negative Symptom Assessment Scale (NSA-16) total score from baseline to endpoint | 16 weeks

SECONDARY OUTCOMES:
Change in the general composite score on the MATRICS Consensus Cognitive Battery (MCCB) from baseline to endpoint | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christoph U Correll, MD, Principal Investigator — North Shore LIJ
Locations (3):
- United States (3):
  - Henderson Behavioral Health, Lauderdale Lakes, Florida
  - Cherry Health, Grand Rapids, Michigan
  - The Zucker Hillside Hospital, Glen Oaks, New York